CLINICAL TRIAL: NCT01133795
Title: Effect of Administration of Intravenous Albumin and Oral Midodrine on Renal Function in Patients With Cirrhosis and Functional Renal Impairment
Brief Title: Midodrine and Albumin for Cirrhotic Patients With Functional Renal Impairment
Acronym: MAFRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Pere Gines, chief of hepatology unit, Hospital Clinic of Barcelona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAFRI
Record Dates: First submitted 2010-05-19; First posted 2010-05-31 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Cirrhosis; Renal Failure
Keywords: cirrhosis; renal failure; hepatorenal syndrome; albumine; midodrine
MeSH Terms: conditions — Fibrosis; Renal Insufficiency; Hepatorenal Syndrome | interventions — Midodrine; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midodrine, Albumin (Experimental): Midodrine 10mg tid for 12 weeks. Albumin 40g every 14 days for 12 weeks
  Interventions: Drug: Midodrine plus Albumin

INTERVENTIONS:
Drug: Midodrine plus Albumin — MIdodrine 10mg tid for 12 weeks. Albumin 40g every 14 days for 12 weeks
  Other Names: Albumin Grifols; Gutron

SUMMARY:
The objective of the study was evaluate the effect of administration of midodrine and albumin on renal function in patients with cirrhosis and creatinine greater than 1,2mg/dl.

DETAILED DESCRIPTION:
Twenty patients with cirrhosis and functional renal impairment, defined by a serum creatinine greater than 1,2mg/dl, will be included. Patients will receive daily midodrine at a dose of 10mg tid and 40g of albumin at 15-day interval. The follow-up period will be of 12 weeks. In all patients, liver and renal function, and vasoactive hormones (plasma renin activity, aldosterone, noradrenaline, ADH, endothelin and anf)will be determined at baseline conditions. At this moment, glomerular filtration rate and renal plasma flow determined by isotopic techniques as ambulatory blood pressure monitoring through a 24-hour period will be performed too. All these determinations will be repeated at 4 and 12 weeks. During the study period, just before the albumin infusions, blood will be drawn for creatinine and electrolytes determinations and these will be recorded as well physical examination performed.

ELIGIBILITY:
Inclusion Criteria:

* Liver Cirrhosis
* Serum Creatinine greater than 1,2 mg/dL
* to have given written informed consent

Exclusion Criteria:

* pregnancy
* Systolic blood pressure above 150mmHg and/or diastolic blood pressure above 90mmHg
* Previous treatment with transjugular intrahepatic portosystemic shunt (TIPS) or surgical shunts
* Antibiotic treatment in the previous 7 days before inclusion, except for prophylaxis of spontaneous bacterial peritonitis
* infection by HIV
* contraindications for albumin and/or midodrine use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in glomerular filtration rate assessed by isotopic methods | at 12 weeks of treatment

SECONDARY OUTCOMES:
changes in arterial pressure as assessed by continuous ambulatory arterial pressure | at 12 weeks of treatment
changes in plasma renin activity | at 12 weeks of treatment
changes in aldosterone concentration | at 12 weeks of treatment
changes in norepinephrine concentration | at 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pere Ginès, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Villarroel 170,Barcelona, Barcelona, Spain